CLINICAL TRIAL: NCT04603001
Title: A Phase 1 Study of Oral LY3410738 in Patients With Advanced Hematologic Malignancies With IDH1 or IDH2 Mutations
Brief Title: Study of Oral LY3410738 in Patients With Advanced Hematologic Malignancies With IDH1 or IDH2 Mutations
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18076; 2020-002830-33 (EudraCT Number); I9Y-OX-JDHB (Other: Eli Lilly and Company); LOXO-IDH-20001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-10-12; First posted 2020-10-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Chronic Myelomonocytic Leukemia (CMML); Myeloproliferative Neoplasms (MPNs)
Keywords: Loxo; LY3410738; isocitrate dehydrogenase; IDH; IDH1; IDH2; R132; R140; R172; 2-hydroxyglutarate; 2-HG; Advanced Hematologic Malignancies; Blasts; Acute Myeloid Leukemia; AML; Relapsed/refractory AML; R/R AML; Myelodysplastic Syndrome; MDS; Chronic Myelomonocytic Leukemia; CMML; Myeloproliferative Neoplasms; MPN; Advanced Hematologic Cancers; Ivosidenib; AG-120; Vorasidenib; AG-881; Olutasidenib; FT-2102; BAY1436032; DS-1001; IDH-305; Enasidenib; AG-221; Arginine 132; Arginine 140; Arginine 172
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation Arm A (Monotherapy) (Experimental): Patients not requiring a strong cytochrome P450 3A4 (CYP3A4) inhibitor.
  Interventions: Drug: LY3410738
- Dose Escalation Arm B (Monotherapy) (Experimental): Patients requiring a strong CYP3A4 inhibitor for active management or prevention of a lifethreatening condition, such as an azole administered to prevent invasive fungal infection.
  Interventions: Drug: LY3410738
- Dose Escalation Arm C (LY3410738, Venetoclax, and Azacitidine) (Experimental): Patients with no prior venetoclax therapy and not requiring a strong CYP3A4 inhibitor for active treatment within 7 days of starting LY3410738.
  Interventions: Drug: LY3410738; Drug: Venetoclax; Drug: Azacitidine
- Cohort 1 (Experimental): Patients with relapsed/refractory (R/R) AML harboring an IDH1 R132 mutation who have received a prior IDH inhibitor.
  Interventions: Drug: LY3410738
- Cohort 2 (Experimental): Patients with R/R AML harboring an IDH1 R132 mutation who have not received a prior IDH inhibitor.
  Interventions: Drug: LY3410738
- Cohort 3 (Experimental): Patients with R/R MDS, chronic myelomonocytic leukemia (CMML) or other advanced hematologic malignancy harboring an IDH1 R132 mutation.
  Interventions: Drug: LY3410738
- Cohort 4 (Experimental): Patients with R/R AML, MDS, CMML or other advanced hematologic malignancy harboring IDH2 mutations.
  Interventions: Drug: LY3410738
- Cohort 5 (Experimental): Patients with newly diagnosed AML, R/R AML, or other advanced hematologic malignancy harboring IDH1 and/or IDH2 mutations with no prior venetoclax therapy. Strong CYP3A4 inhibitor allowed but not required.
  Interventions: Drug: LY3410738; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: LY3410738 — Oral LY3410738
Drug: Venetoclax — Oral venetoclax
  Arms: Cohort 5; Dose Escalation Arm C (LY3410738, Venetoclax, and Azacitidine)
Drug: Azacitidine — Subcutaneous or intravenous azacitidine
  Arms: Cohort 5; Dose Escalation Arm C (LY3410738, Venetoclax, and Azacitidine)

SUMMARY:
This is an open-label, multi-center Phase 1 study of LY3410738, an oral, covalent isocitrate dehydrogenase (IDH) inhibitor, in patients with IDH1 and/or IDH2-mutant advanced hematologic malignancies who may have received standard therapy

DETAILED DESCRIPTION:
This study includes 2 parts: dose escalation and dose expansion. The dose escalation will enroll eligible patients with select IDH-mutant advanced hematologic malignancies. Once the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of LY3410738 is established, the dose expansion will begin and enroll into 5 cohorts to further evaluate safety and clinical activity

ELIGIBILITY:
Inclusion Criteria:

* Advanced IDH mutant hematologic malignancy including:

  -- For Dose Escalation Arm C and Dose Expansion Cohort 5:
  * Patients with newly diagnosed AML who are 75 years or older or have comorbidities that preclude the use of intensive chemotherapy
  * Patients with R/R AML (US only)
* Patients must have received prior therapy
* Blasts at least 5% in bone marrow.
* Patients must have a qualifying IDH1 R132, IDH2 R140 or IDH2 R172 mutation
* Eastern Cooperative Oncology Group (ECOG) 0 to 2
* Adequate organ function
* Ability to swallow capsules or tablets
* Ability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation
* Willingness of men and women of reproductive potential to observe conventional and effective birth control for the duration of treatment and for 3 months following the last dose of study treatment.

Exclusion Criteria:

* Investigational agent or anticancer therapy within 2 weeks or 5 half-lives, whichever is shorter; or investigational monoclonal antibody within 4 weeks prior to planned start of LY3410738
* For Dose Escalation Arm C and Dose Expansion Cohort 5:

  * Prior venetoclax treatment is not allowed.
  * Patients are allowed to receive up to 1 cycle of single agent azacitidine or azacitidine plus venetoclax while waiting for results of locally obtained molecular profiling, including IDH1/IDH2 mutational status, prior to starting on study.
* Major surgery within 4 weeks prior to planned start of LY3410738.
* Active, uncontrolled clinically significant systemic bacterial, viral, fungal or parasitic infection or an unexplained fever > 38.5ºC during Screening or on the first day of study drug administration.
* Another concurrent malignancy requiring active therapy.
* Active central nervous system involvement
* Any unresolved toxicities from prior therapy greater than CTCAE v5.0 Grade 2 at the time of starting study treatment except for alopecia.
* History of hematopoietic stem cell transplant (HSCT) or chimeric antigen receptor T-cell (CAR-T) therapy within 60 days of the first dose of LY3410738.
* Clinically significant cardiovascular disease
* Active hepatitis B virus (HBV)
* Active hepatitis C virus (HCV)
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of the study drug
* Current treatment with certain strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers and/or P- glycoprotein (P-gp) inhibitor, with the exception of patients being treated with allowed antifungal inhibitors of CYP3A4
* Treatment with proton pump inhibitor (PPIs) within 7 days of starting LY3410738
* Any serious underlying medical or psychiatric condition (e.g. alcohol or drug abuse), dementia or altered mental status or any issue that would impair the ability of the patient to understand informed consent or that in the opinion of the Investigator would contraindicate the patient's participation in the study or confound the results of the study
* Known human immunodeficiency virus (HIV), excluded due to potential drug-drug interactions between antiretroviral medications and LY3410738
* Pregnancy, lactation or plan to breastfeeding during the study or within 90 days of the last dose of study intervention
* Known hypersensitivity to any of the components of LY3410738 or its formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) | Up to 30 months
  For Dose Escalation
To assess the activity of LY3410738 as measured by the overall response rate (ORR) per the Investigator assessment | Up to 30 months
  For Dose Expansion

SECONDARY OUTCOMES:
To determine the safety profile and tolerability of LY3410738 including acute and chronic toxicities by collecting and evaluating adverse events and treatment emergent adverse events | Up to 30 months
  For Dose Escalation
To characterize the pharmacokinetics (PK) properties of LY3410738 by collecting and evaluating serum at protocol specified time points | Up to 30 months
  For Dose Escalation
To characterize the pharmacodynamic properties of LY3410738 as expressed by change in 2-HG oncometabolite levels in plasma | Up to 30 months
  For Dose Escalation
To assess the activity of LY3410738 as measured by the overall response rate (ORR) per Investigator assessment | Up to 30 months
  For Dose Escalation
To assess the activity of LY3410738 as measured by Best Overall Response (BOR) per Investigator assessment | Up to 30 months
  For Dose Expansion
To assess the activity of LY3410738 by Complete Remission (CR) Rate (CRR) plus partial hematologic recovery (AML patients) | Up to 30 months
  For Dose Expansion
To assess the activity of LY3410738 by Duration of Response | Up to 30 months
  For Dose Expansion
To assess the activity of LY3410738 by Hematologic improvement in patients with MDS | Up to 30 months
  For Dose Expansion
To determine the safety profile and tolerability of LY3410738 including acute and chronic toxicities by collecting and evaluating Adverse events and treatment emergent adverse events | Up to 30 months
  For Dose Expansion
To characterize the pharmacokinetics (PK) properties of LY3410738 by collecting and evaluating serum at protocol specified time points | Up to 30 months
  For Dose Expansion
To characterize the pharmacodynamic properties of LY3410738 as expressed by change in 2-HG oncometabolite levels in plasma. | Up to 30 months
  For Dose Expansion

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (12):
  - City of Hope National Medical Center, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - University of California, Davis - Health Systems, Sacramento, California
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- Canada (3):
  - BC Cancer Vancouver, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus), Helsinki, Finland
- France (5):
  - Institut Paoli-Calmettes, Marseille
  - Hopital Saint Louis, Paris
  - Centre hospitalier universitaire de Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Claudius Regaud, Toulouse
- Medizinische Hochschule Hanover, Hanover, Lower Saxony, Germany
- Rambam Medical Center, Haifa, Israel
- Singapore (2):
  - National University Cancer Institute, Singapore
  - Singapore General Hospital, Singapore
- South Korea (3):
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Seoul National University Hospital, Seoul
- Spain (3):
  - Clinico Y Provincial Barcelona, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Fe de Valencia, Valencia
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study of LY3410738 in Patients with Advanced Blood Cancers with a Change in the IDH1 or IDH2 Gene — https://trials.lillytrialguide.com/en-US/trial/5zLVhd8jkDNg8KcTGH3Tf9?nickname=I9Y-OX-JDHB